CLINICAL TRIAL: NCT05502679
Title: Immediate Versus Late Weight Bearing After Tibial Plateau Fractures Internal Fixation: A Randomized Clinical Trial
Brief Title: Immediate Versus Late Weight Bearing After Tibial Plateau Fractures Internal Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Texas Tech University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Mariam ibrahim, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17200756
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Fracture of Tibia Proximal Plateau
Keywords: rehabilitation; radiography; physical therapy; intra-articular knee fracture
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Weight-Bearing

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The first patient from each type of Schatzker classification 1-4 tibial plateau fractures will be randomly assigned to either WBG or TG. Then each patient will be alternatively assigned to WBG or TG as a stratification method to ensure that each group has equal distribution from each type of Schatzker classification 1-4 tibial plateau fractures. The randomization file will be generated by an investigator (TH) not involved in the data collection process, with the results stored in a spreadsheet accessible only to the investigator responsible for the subjects' group assignment (MI). This investigator will not participate in any data collection or subject treatment. Due to the nature of the study, participants will not be blinded to the group assignment and treatment they will receive. However, the investigators measuring the dependent variables will be blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Group (Active Comparator): 6-week non-weight bearing of the affected lower limb rehabilitation protocol (TG)
  Interventions: Other: Pragmatic Exercise protocol
- Weight-bearing Group (Experimental): Immediate lower limb weight bearing to tolerance rehabilitation protocol (WBG)
  Interventions: Other: Weight bearing as tolerated; Other: Pragmatic Exercise protocol

INTERVENTIONS:
Other: Weight bearing as tolerated — Bearing weight on lower limb extremity
  Arms: Weight-bearing Group
Other: Pragmatic Exercise protocol — Designed exercise prescriptions according to the patients' needs

SUMMARY:
Postoperative rehabilitation for tibial plateau fracture generally involves prolonged non-weight bearing time while other protocols use partial weight-bearing and bracing before full weight-bearing is recommended at 9 to 12 weeks following surgical fixation. No study to date has investigated the effect of standardized pragmatic exercise protocol added to immediate weight bearing after tibial plateau fractures surgical fixation on patient's functional outcomes, knee ROM, pain, radiographic boney alignment, gait, and return to work.

DETAILED DESCRIPTION:
Tibial plateau fractures can permanently affect patients' quality of life, including significant socio-economic impact due to time off work, compromised knee functional integrity, secondary knee osteoarthritis, knee flexion contractures, job loss due to functional limitations, and limited ability to return to pre-injury level of sports participation. Additionally, patients with tibial plateau fracture are at greater risk of death compared to an age- and the gender-matched reference population.

In orthopedics, weight-bearing refers to how much weight a person bears through an injured body part. During a single-leg stance, a person with no physical limitations will carry 100% of their body weight through each leg. Thus, grades of weight bearing are generally expressed as a percent of the body weight. Weight-bearing grades include (1) Non-weight bearing (NWB), which means the patient is not to put any weight through the affected limb(s); (2) Toe touch weight bearing (TTWB), which is poorly defined in the literature. In clinical practice, it is commonly described as having the ability to touch the toes to the floor without supporting weight from the affected limb. The pressure should be light enough to avoid crushing a potato crisp underfoot. Partial weight bearing (PWB) can range from anything greater than non-weight bearing to anything less than full weight bearing. The status is usually accompanied by a percentage figure to describe the extent of recommended weight bearing further. Most of the definitions in the literature define partial weight bearing as being 30% to 50% of a patient's body weight. Full weight bearing (FWB) means no restriction to weight bearing. In other words, 100% of a person's body weight can be transmitted through the designated limb. This term is somewhat interchangeable with the term 'weight bear as tolerated (WBAT), which allows them to self-limit their weight bearing up to full body weight. Restriction in weight bearing of the operated leg during standing and walking is needed to avoid complications during the postoperative recovery such as mal-union, fracture reduction loss, or hardware failure.

Postoperative rehabilitation for tibial plateau fracture generally involves prolonged non-weight bearing time, while other protocols use partial weight-bearing and bracing before full weight-bearing is recommended at 9 to 12 weeks following fixation. Early weight-bearing and early range of motion (ROM) for cartilage nourishment and preservation after selected lower limb surgical procedures are associated with positive postoperative outcomes, including decreased mortality and morbidity rate, functional improvements, reduced inpatient length of stay, and improved healing process. Early weight-bearing prescription, however, has to be carefully assessed, as it may result in fracture reduction loss, hardware failure, infection, malunion, or nonunion. The effectiveness of immediate partial post-operative weight-bearing in the management of lateral tibial plateau fractures resulted in favorable outcomes after immediate partial weight-bearing of 15 kg in cases of bicondylar tibial plateau fractures fixed with medial and lateral plating, and after immediate partial weight-bearing, up to 25 kg in all types of tibial plateau fractures fixed using a range of approaches.

By using locking plates for tibial plateau fracture surgical management, surgeons can safely allow immediate postoperative weight-bearing. Immediate weight bearing did not produce additional tibial plateau depression greater than 2 mm with Schatzker Type I, II, III, or Type V fractures. This could potentially reduce the rate of postoperative complications due to immobilization, such as deep venous thrombosis and joint stiffness.

Knee ROM limitations and altered gait characteristics are common complications after tibial plateau fractures. Most gait improvements occurred within the first postoperative six months. The total ROM at each lower limb joint showed positive correlations with the patients' capability to conduct normal activities of daily living.

To the authors' knowledge, no randomized control study to date has investigated in patients following tibial plateau fracture surgical fixation the effect of (1) adding immediate weight bearing to tolerance in addition to a specific, tailored exercise program adapted to the type and mechanism of tibial plateau fractures; and (2) adding phones follow-ups to improve compliance and decrease the cost of care.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men (18 to 65 years of age) admitted to Assiut University Hospital - Trauma unit with the diagnosis of traumatic tibial plateau closed fracture.
2. Open or arthroscopic internal fixation for tibial plateau fracture.
3. Schatzker classification 1-4 tibial plateau fractures.
4. An Orthopedic surgeon with at least 5 years of surgery experience.
5. Precontoured and standard locking compression plates for the tibia plateau fracture internal fixation.

Exclusion Criteria:

1-. Contralateral limb condition that prevents weight-bearing 3. Ipsilateral injuries such as tibial or femoral fractures, hip fractures, or pelvic ring injuries.

4. Patients are required to wear a locking knee brace following the surgical fixation for a concomitant ligamentous knee injury.

5. Patient treated conservatively or with external fixation. 6. Surgical fixation is delayed for more than 10 days after the injury. 7. Requirement of involved leg fixed immobilization (e.g., cast) following the surgical fixation 8. Non-ambulatory pre-tibial plateau fracture 9. Pre-injury limitation to ROM of ipsilateral knee 10. Documented psychiatric disorder (aggressive, bipolar) requiring admission in the perioperative period.

11. Cognitive or mental condition that prevents the patient from following directions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
The change in Oxford knee score (OKS) from 6 weeks to 3 months and 6 months after surgery | 6 weeks, 3 and 6 months after the surgery
  Arabic version of Oxford knee score.Functional knee questionnaire.The questionnaire consists of 12 questions that cover the function and pain of the knee. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes.
The change in active Knee range of motion | Baseline, 2 and 6 weeks, 3months after the surgery
  Measuring Active knee flexion and extension and at 3 month tibial rotation ROM will be measured
The change of radiograph measurements on X-ray | Baseline and 3 months after the surgery
  proximal medial tibial angle to detect varus / valgus angulation .
The change on clinical impression of reduction quality on Computed tomography | Baseline and 3 months after the surgery
  measurement of fracture gap, joint step off, tibial plateau width, tibial slope and depression will be measured to report quality of reduction and bony alignment.

SECONDARY OUTCOMES:
Return to work Assessment | 3- and 6-month post-surgery
  Time to return to work and either return to the same job or not
The change in Hip Stability Isometric Tests and knee extensor strength using (handheld dynamometer) | 6 weeks and 3 months after the surgery
  measuring the isometric muscle strength

OTHER OUTCOMES:
Satisfaction with weight bearing protocol | 3 month after the surgery
  yes or no question
The change in average pain intensity of the lower leg using the numeric Pain Rating Scale | Baseline, 2 and 6 weeks, 3 and 6 months after surgery
  Scores range from 0-10 points, with higher scores indicating greater pain intensity.
Anatomical relationship of articular surfaces on X-ray | 6 weeks after surgery
  Redflags regarding Articular congruency,the anatomical relationship of articular surfaces with or without hardware failure (Yes / NO) and visual intra-articular collapse will be measured to report bone alignment quality on x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Brismee, Professor, Study Chair — Texas Tech Health Sciences Center
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available for the other researchers and reviewers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 30 days
Access Criteria: Via email

REFERENCES:
- [Background] Ahmed KM, Said HG, Ramadan EKA, Abd El-Radi M, El-Assal MA. Arabic translation and validation of three knee scores, Lysholm Knee Score (LKS), Oxford Knee Score (OKS), and International Knee Documentation Committee Subjective Knee Form (IKDC). SICOT J. 2019;5:6. doi: 10.1051/sicotj/2018054. Epub 2019 Mar 8. PMID 30848244